CLINICAL TRIAL: NCT00704262
Title: Effect of Calcipotriol Plus Hydrocortisone Ointment on the Hypothalamic-pituitary-adrenal (HPA) Axis and Calcium Metabolism in Patients With Psoriasis Vulgaris on the Face and on the Intertriginous Areas
Brief Title: Effect of Calcipotriol Plus Hydrocortisone Ointment on the Adrenal Hormone Balance and Calcium Metabolism in Patients With Psoriasis Vulgaris on the Face and Skin Folds
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEO 80190-O23
Record Dates: First submitted 2008-06-23; First posted 2008-06-24 (Estimated); Results first posted 2020-10-20 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2020-09

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — calcipotriene; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Calcipotriol plus hydrocortisone (LEO 80190) (Experimental)
  Interventions: Drug: Calcipotriol plus hydrocortisone (LEO 80190)

INTERVENTIONS:
Drug: Calcipotriol plus hydrocortisone (LEO 80190) — Once daily application

SUMMARY:
There are few therapies suitable for the treatment of psoriasis on the face and skin folds. As these areas are sensitive, irritation and other adverse reactions are more common than elsewhere on the body. The purpose of the study is to monitor the effect of once daily treatment for up to 8 weeks of an ointment containing calcipotriol 25 mcg/g plus hydrocortisone 10 mg/g on the hypothalamic-pituitary-adrenal axis and on the calcium metabolism in patients with psoriasis vulgaris on the face and on the intertriginous areas

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of psoriasis vulgaris involving the face and the intertriginous areas
* Clinical diagnosis of psoriasis vulgaris on the trunk and/or limbs or earlier diagnosed with psoriasis vulgaris on the trunk and/or limbs
* An extent of psoriatic involvement on the face of at least 5 cm2 and the sum of all facial and intertriginous lesions at least 30 cm2
* Treatment areas (face and intertriginous) amenable to topical treatment with a maximum of 100g ointment per week
* Disease severity of the face and intertriginous areas graded as moderate, severe or very severe according to the investigator´s global assessment of disease severity
* Patients with a normal HPA axis function: serum cortisol concentration above 5 mcg/dl before adrenocorticotropic hormone (ACTH: tetracosactid/cosyntropin) injection and serum cortisol concentration above 18 mcg/dl 30 min after ACTH (tetracosactid/cosyntropin) injection
* Albumin corrected serum calcium within reference range
* Females of childbearing potential have to use a highly effective method of contraception during the study (hormonal contraceptives on oestrogen basis are not allowed)

Exclusion Criteria:

* A history of active allergy, asthma, allergic skin rash, or sensitivity to any medication (including ACTH/tetracosactid/cosyntropin) or to any component of the formulations being tested
* Systemic treatment with all other therapies than biologicals, with a potential effect on psoriasis vulgaris (eg vitamin D analogues, retinoids)within 2 weeks prior to Visit 1. Stable treatment with methotrexate or fumaric acid is allowed
* Systemic treatment with corticosteroids within 12 weeks prior to Visit 1
* Systemic use of biological treatments, whether marketed or not, directed against or with a potential effect on psoriasis vulgaris (eg. alefacept, efalizumab, etanercept, infliximab, adalimumab) within 12 weeks prior to Visit 1
* Psoralen plus ultraviolet light A (PUVA) therapy or Grenz ray therapy within 4 weeks prior to Visit 1
* Ultraviolet B (UVB) therapy within 2 weeks prior to Visit 1
* Topical treatment with World Health Organization (WHO) group 2, 3 or 4 corticosteroids within 4 weeks prior to Visit 1
* Topical treatment with WHO group 1 corticosteroids within 2 weeks prior to Visit 1
* Any topical treatment of the face and intertriginous areas (except for emollients) within 2 weeks prior to Visit 1
* Oestrogen therapy or any other medication known to affect cortisol levels or HPA-axis integrity within 4 weeks prior to Visit 1
* Enzymatic inductors, systemic or topical cytochrome P450 inhibitors, hypoglycaemic sulfonamides or antidepressive medication within 4 weeks prior to Visit 1
* Current diagnosis of erythrodermic, exfoliative, guttate or pustular psoriasis
* Patients with any of the following conditions present on the treatment area: viral (e.g., herpes or varicella) lesions of the skin, fungal and bacterial skin infections, parasitic infections, skin manifestations in relation to syphilis or tuberculosis, rosacea, perioral dermatitis, acne vulgaris, atrophic skin, striae atrophicae, fragility of skin veins, ichthyosis, acne rosacea, ulcers and wounds
* Other inflammatory skin diseases (e.g., seborrhoeic dermatitis, contact dermatitis and cutaneous mycosis) that may confound the evaluation of psoriasis vulgaris on the face or on the intertriginous areas
* Planned exposure to sun, Ultraviolet A (UVA) or UVB during the study that may affect the psoriasis vulgaris
* Clinical signs or symptoms of Cushing´s disease or Addison's disease
* Known or suspected severe renal insufficiency or severe hepatic disorders
* Known or suspected disorders of calcium metabolism associated with hypercalcaemia
* Known or suspected endocrine disorder that may affect the results of the ACTH challenge test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rainard Fuhr, MD, PhD, Principal Investigator — Institute of Pharmacology Parexel International GmbH, Spandauer Damm 130, Haus 31, 14050 Berlin, Germany
Locations (11):
- United States (6):
  - Burke Pharmaceuticals, Hot Springs, Arkansas
  - Dermatology Research of Arkansas, Little Rock, Arkansas
  - Ameriderm Research, Ormond Beach, Florida
  - Somerset Skin Center, Troy, Michigan
  - Psoriasis Treatment Center of Central NJ, East Windsor, New Jersey
  - Virginia Clinical Research, Inc., Norfolk, Virginia
- The Guenther Dermatology Research Centre, London, Ontario, Canada
- Institute of Clinical Pharmacology Parexel International Gmbh, Berlin, Germany
- United Kingdom (3):
  - LCG Bioscience, Bourn, Cambridge
  - ICON Development Solutions, Manchester
  - The Dermatology Centre, Hope Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The treatment phase was divided into two 4-week treatment periods during which the overall treatment duration had to be 28 days or 56 days. The participant was to leave the study if they were clear according to the investigator's global assessment of disease severity (IGA) of the face and of the intertriginous areas at Visit 3 (Day 28).
Groups:
- Calcipotriol Plus Hydrocortisone (LEO 80190): Calcipotriol plus hydrocortisone (LEO 80190) ointment applied topically once daily for either 28 or 56 consecutive days on psoriasis vulgaris affected skin on the face and on the intertriginous areas.
  The ointment was not to be applied in the 24-hour period before Day 28 and Day 56 to avoid interference from the hydrocortisone with the adrenocorticotrophic hormone (ACTH) challenge test. Treatment was to be resumed after Visit 3, where applicable.
  The face was defined as: forehead including hairline, cheeks, nose, chin and ears (excluding the auditory meatus). In case of baldness or partial baldness, the forehead was to be estimated considering the standard or previous hairline. The intertriginous areas were defined as the axillae, the genito-femoral and inguinal folds, the inframammary folds, the intergluteal folds, and scrotum.
Period: Overall Study
Arm/Group | Calcipotriol Plus Hydrocortisone (LEO 80190)
Started | 33
Completed | 31
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Calcipotriol Plus Hydrocortisone (LEO 80190)
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 19
Region of Enrollment [Number; unit: participants]
  Canada | 8
  United States | 7
  United Kingdom | 11
  Germany | 7

OUTCOME MEASURES:

1. Primary Outcome: The Adrenal Response to the ACTH Challenge Test Defined as the Serum Cortisol Concentration Obtained After 30 and 60 Minutes
Description: The adrenal function was assessed by a rapid standard dose ACTH (tetracosactid/cosyntropin) challenge test. The ACTH challenge test consisted of a baseline blood (Day -7 to Day -3) sample taken at 8 a.m. (± 30 minutes). Following the baseline blood sample, an intravenous bolus injection of 250 mcg Synacthen®/Cortrosyn® was given at Time 0 (T = 0). Serum cortisol concentrations at 30 and 60 minutes after administration were taken and reflected the stimulation induced by tetracosactid/cosyntropin.
  ≤18 mcg/dL was considered low.
Time Frame: At Week 4 (Day 28) and Week 8 (Day 56)
Population: Per protocol analysis set (out of 33 participants who received treatment, 1 provided no ACTH challenge test data following start of treatment and 2 applied less than 1 gram of study treatment.)
Measure: Count of Participants; unit: Participants
Arm/Group | Calcipotriol Plus Hydrocortisone (LEO 80190)
Number analyzed (Participants) | 30
Participants
  >18 mcg/dL | 29
  ≤18 mcg/dL | 1

2. Primary Outcome: Change in Albumin Corrected Serum Calcium
Description: Baseline was defined as the last assessment performed before study medication application. The end of treatment data was defined as the last value recorded during the treatment phase (i.e. Week 4, 6, or 8).
Time Frame: From baseline to Week 4, Week 8, and end of treatment (last value recorded i.e. Week 4, 6, or 8)
Population: This evaluation was based on the safety analysis set that consists of all participants who received at least one application with study treatment (33 participants). The analysis only contains data from participants who attended the specific visits.
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Calcipotriol Plus Hydrocortisone (LEO 80190)
Number analyzed (Participants) | 33
mmol/L
  Baseline | 2.215 [2.188 to 2.243]
  Week 4 (Day 28) | 0.002 [-0.026 to 0.029]
  Week 8 (Day 56): number analyzed (Participants) | 27
  Week 8 (Day 56) | -0.045 [-0.083 to -0.007]
  End of Treatment (last value recorded) | -0.033 [-0.066 to 0.000]

3. Secondary Outcome: The Adrenal Response to the ACTH Challenge Test Defined as the Serum Cortisol Concentration Obtained After 30 Minutes
Description: as for outcome 1
Time Frame: At Week 4 and Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Calcipotriol Plus Hydrocortisone (LEO 80190)
Number analyzed (Participants) | 30
Participants
  >18 mcg/dL | 29
  ≤18 mcg/dL | 1

4. Secondary Outcome: The Adrenal Response to the ACTH Challenge Test Defined as the Serum Cortisol Concentration Obtained After 60 Minutes
Description: as for outcome 1
Time Frame: At Week 4 and Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Calcipotriol Plus Hydrocortisone (LEO 80190)
Number analyzed (Participants) | 30
Participants
  >18 mcg/dL | 30
  ≤18 mcg/dL | 0

5. Secondary Outcome: Serum Cortisol Concentration After 30 Minutes
Description: The adrenal function was assessed by a rapid standard dose ACTH (tetracosactid/cosyntropin) challenge test. The ACTH challenge test consisted of a baseline blood (Day -7 to Day -3) sample taken at 8 a.m. (± 30 minutes). Following the baseline blood sample, an intravenous bolus injection of 250 mcg Synacthen®/Cortrosyn® was given at Time 0 (T = 0). Serum cortisol concentrations at 30 and 60 minutes after administration were taken and reflected the stimulation induced by tetracosactid/cosyntropin.
Time Frame: At Week 4 and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | Calcipotriol Plus Hydrocortisone (LEO 80190)
Number analyzed (Participants) | 30
mcg/dL
  Week 4 (Day 28) | 25.29 (4.35)
  Week 8 (Day 56): number analyzed (Participants) | 26
  Week 8 (Day 56) | 25.93 (4.73)

6. Secondary Outcome: Serum Cortisol Concentration After 60 Minutes
Description: as for outcome 5
Time Frame: At Week 4 and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | Calcipotriol Plus Hydrocortisone (LEO 80190)
Number analyzed (Participants) | 30
mcg/dL
  Week 4 (Day 28) | 28.81 (3.48)
  Week 8 (Day 56): number analyzed (Participants) | 27
  Week 8 (Day 56) | 28.82 (5.30)

7. Secondary Outcome: Change in Albumin Corrected Serum Calcium
Description: Baseline was defined as the last assessment performed before study medication application.
Time Frame: From baseline to Week 2 and Week 6
Population: This evaluation was based on all participants who received at least one application with study treatments, thus 33 participants were analyzed. The table only contains data from participants who attended the specific visits.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Calcipotriol Plus Hydrocortisone (LEO 80190)
Number analyzed (Participants) | 33
mmol/L
  Baseline | 2.215 (0.077)
  Week 2 (Day 14): number analyzed (Participants) | 32
  Week 2 (Day 14) | 0.018 (0.095)
  Week 6 (Day 42): number analyzed (Participants) | 28
  Week 6 (Day 42) | -0.013 (0.083)

8. Secondary Outcome: Albumin Corrected Serum Calcium
Description: The end of treatment data was defined as the last value recorded during the treatment phase (i.e. Week 4, 6, or 8).
Time Frame: At Week 2, Week 4, Week 6 and Week 8 and end of treatment (last value recorded i.e. Week 4, 6, or 8)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Calcipotriol Plus Hydrocortisone (LEO 80190)
Number analyzed (Participants) | 33
mmol/L
  Week 2 (Day 14): number analyzed (Participants) | 32
  Week 2 (Day 14) | 2.233 (0.079)
  Week 4 (Day 28) | 2.217 (0.074)
  Week 6 (Day 42): number analyzed (Participants) | 28
  Week 6 (Day 42) | 2.208 (0.096)
  Week 8 (Day 56): number analyzed (Participants) | 27
  Week 8 (Day 56) | 2.179 (0.085)
  End of Treatment (last value recorded) | 2.182 (0.081)

9. Secondary Outcome: Albumin Corrected Serum Calcium Values Above the Upper Limit of the Reference Range
Description: The table summarizes the shifts in albumin corrected serum calcium versus the normal range. The end of treatment data was defined as the last value recorded for the parameter during the treatment phase of the study (i.e. Week 4, 6, or 8).
  The normal reference range for the albumin corrected serum calcium was defined as 2.1-2.64 mmol/L (8.4-10.6 mg/L). The value below this level was considered 'low', while the value above this range was considered 'high'.
Time Frame: At Week 2, Week 4, Week 6 and Week 8 and end of treatment (last value recorded i.e. Week 4, 6, or 8)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Calcipotriol Plus Hydrocortisone (LEO 80190)
Number analyzed (Participants) | 33
Participants
  Week 2 (Day 14): number analyzed (Participants) | 32
  Week 2 (Day 14): Low | 2
  Week 2 (Day 14): Normal | 30
  Week 2 (Day 14): High | 0
  Week 4 (Day 28): Low | 3
  Week 4 (Day 28): Normal | 30
  Week 4 (Day 28): High | 0
  Week 6 (Day 42): number analyzed (Participants) | 28
  Week 6 (Day 42): Low | 2
  Week 6 (Day 42): Normal | 26
  Week 6 (Day 42): High | 0
  Week 8 (Day 56): number analyzed (Participants) | 27
  Week 8 (Day 56): Low | 6
  Week 8 (Day 56): Normal | 21
  Week 8 (Day 56): High | 0
  End of Treatment (last value recorded): Low | 6
  End of Treatment (last value recorded): Normal | 27
  End of Treatment (last value recorded): High | 0

10. Secondary Outcome: Participants With "Controlled Disease" ("Clear" or "Almost Clear") According to the Investigator's Global Assessment of Disease Severity (IGA) of the Face
Description: Controlled disease was defined as the following (P=Plaque thickening, S=Scaling, E=Erythema) Clear (Plaque thickening=no elevation/thickening of normal skin, S=no evidence of scaling, E= none/hyperpigmentation/residual red coloration) or Almost clear (P=none/possible thickening but difficult to ascertain whether there is a slight elevation above normal skin level, S=none/residual surface dryness and scaling, E=light pink coloration) (last value recorded i.e. Week 4, 6, or 8)
Time Frame: At Week 4, Week 8 and end of treatment (last value recorded i.e. Week 4, 6, or 8)
Population: This efficacy evaluation is based on the full analysis set that consists of all participants who received study treatment, thus 33 participants were analyzed. The analysis only contains data from participants who attended the specific visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Calcipotriol Plus Hydrocortisone (LEO 80190)
Number analyzed (Participants) | 33
Participants
  Week 4 (Day 28): Controlled | 21
  Week 4 (Day 28): Non-controlled | 12
  Week 8 (Day 56): number analyzed (Participants) | 28
  Week 8 (Day 56): Controlled | 19
  Week 8 (Day 56): Non-controlled | 9
  End of Treatment (last value recorded): Controlled | 23
  End of Treatment (last value recorded): Non-controlled | 10

11. Secondary Outcome: Participants With "Controlled Disease" ("Clear" or "Almost Clear") According to the IGA of the Intertriginous Areas
Description: Controlled disease was defined as the following:
  Clear (Infiltration = no elevation or thickening of normal skin, Erythema = normal skin colour or hyperpigmentation) or Almost clear (Infiltration = no elevation or thickening of normal skin, Erythema = faint pink colour) The end of treatment data was defined as the last value recorded for the efficacy measure.
Time Frame: At Week 4, Week 8 and end of treatment (last value recorded i.e. Week 4, 6, or 8)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Calcipotriol Plus Hydrocortisone (LEO 80190)
Number analyzed (Participants) | 33
Participants
  Week 4 (Day 28): Controlled | 20
  Week 4 (Day 28): Non-controlled | 13
  Week 8 (Day 56): number analyzed (Participants) | 28
  Week 8 (Day 56): Controlled | 19
  Week 8 (Day 56): Non-controlled | 9
  End of Treatment (last value recorded): Controlled | 23
  End of Treatment (last value recorded): Non-controlled | 10

12. Secondary Outcome: Overall Disease Severity of the Face According to the IGA
Description: 6-category scale based on plaque thickening (P), Scaling (S), Erythema (E). Clear (P=no elevation/thickening of normal skin, S=no evidence of scaling, E=none/hyperpigmentation/residual red coloration) Almost clear (P=none/possible thickening but difficult to ascertain whether there is a slight elevation above normal skin level, S=none/residual surface dryness and scaling, E=light pink coloration) Mild (P=slight but definite elevation, S=fine scales partially/mostly covering lesions, E=light red coloration) Moderate (P=moderate elevation with rounded or sloped edges, S=most lesions at least partially covered, E=definite red coloration) Severe (P =marked elevation typically with hard or sharp edges, S=non-tenacious scale predominates, covering most or all of the lesions, E=very bright red coloration) Very severe (P=very marked elevation typically with hard or sharp edges, S=thick tenacious scale covers most or all of the lesions, E=extreme red coloration, deep red coloration)
Time Frame: At baseline, Week 2, Week 4, Week 6, Week 8, and end of treatment (last value recorded i.e. Week 4, 6, or 8)
Population: A participant was to leave the study if he/she was clear according to the IGA of the face and after 4 weeks of treatment. Participants who still had psoriasis on the face after 4 weeks of treatment continued treatment for another 4-week period.
Measure: Count of Participants; unit: Participants
Arm/Group | Calcipotriol Plus Hydrocortisone (LEO 80190)
Number analyzed (Participants) | 33
Participants
  Baseline: Clear | 0
  Baseline: Almost clear | 0
  Baseline: Mild | 0
  Baseline: Moderate | 27
  Baseline: Severe | 6
  Baseline: Very severe | 0
  Week 2 (Day 14): Clear | 0
  Week 2 (Day 14): Almost clear | 12
  Week 2 (Day 14): Mild | 15
  Week 2 (Day 14): Moderate | 5
  Week 2 (Day 14): Severe | 1
  Week 2 (Day 14): Very severe | 0
  Week 4 (Day 28): Clear | 5
  Week 4 (Day 28): Almost clear | 16
  Week 4 (Day 28): Mild | 9
  Week 4 (Day 28): Moderate | 2
  Week 4 (Day 28): Severe | 1
  Week 4 (Day 28): Very severe | 0
  Week 6 (Day 42): number analyzed (Participants) | 28
  Week 6 (Day 42): Clear | 5
  Week 6 (Day 42): Almost clear | 15
  Week 6 (Day 42): Mild | 7
  Week 6 (Day 42): Moderate | 1
  Week 6 (Day 42): Severe | 0
  Week 6 (Day 42): Very severe | 0
  Week 8 (Day 56): number analyzed (Participants) | 28
  Week 8 (Day 56): Clear | 5
  Week 8 (Day 56): Almost clear | 14
  Week 8 (Day 56): Mild | 6
  Week 8 (Day 56): Moderate | 3
  Week 8 (Day 56): Severe | 0
  Week 8 (Day 56): Very severe | 0
  End of Treatment (last value recorded): Clear | 9
  End of Treatment (last value recorded): Almost clear | 14
  End of Treatment (last value recorded): Mild | 6
  End of Treatment (last value recorded): Moderate | 3
  End of Treatment (last value recorded): Severe | 1
  End of Treatment (last value recorded): Very severe | 0

13. Secondary Outcome: Overall Disease Severity of Intertriginous Areas According to the IGA
Description: The assessment of the disease severity of the intertriginous areas was made using the 6-category scale; clear, almost clear, mild, moderate, severe, very severe.
  Clear (Infiltration = no elevation or thickening of normal skin, Erythema = normal skin colour or hyperpigmentation) Almost clear (Infiltration = no elevation or thickening of normal skin, Erythema = faint pink colour) Mild (Infiltration = slight, subtle thickening or infiltration, only marginally increased from normal skin, Erythema = light pink colour) Moderate (Infiltration = palpable thickening or infiltration without elevation, Erythema = definite pink colour) Severe (Infiltration = palpable thickening or infiltration with elevation, Erythema = very bright red coloration) Very severe (Infiltration = marked thickening or infiltration with rounded or sloped edges, Erythema = bright deep red coloration)
Time Frame: At baseline, Week 2, Week 4, Week 6, Week 8, and end of treatment (last value recorded i.e. Week 4, 6, or 8)
Population: A participant was to leave the study if they were clear according to the IGA of the intertriginous after 4 weeks of treatment. Participants who still had psoriasis on the intertriginous areas after 4 weeks of treatment continued treatment for another 4-week period.
Measure: Count of Participants; unit: Participants
Arm/Group | Calcipotriol Plus Hydrocortisone (LEO 80190)
Number analyzed (Participants) | 33
Participants
  Baseline: Clear | 0
  Baseline: Almost clear | 0
  Baseline: Mild | 0
  Baseline: Moderate | 19
  Baseline: Severe | 12
  Baseline: Very severe | 2
  Week 2 (Day 14): Clear | 0
  Week 2 (Day 14): Almost clear | 7
  Week 2 (Day 14): Mild | 16
  Week 2 (Day 14): Moderate | 9
  Week 2 (Day 14): Severe | 1
  Week 2 (Day 14): Very severe | 0
  Week 4 (Day 28): Clear | 5
  Week 4 (Day 28): Almost clear | 15
  Week 4 (Day 28): Mild | 10
  Week 4 (Day 28): Moderate | 2
  Week 4 (Day 28): Severe | 1
  Week 4 (Day 28): Very severe | 0
  Week 6 (Day 42): number analyzed (Participants) | 28
  Week 6 (Day 42): Clear | 4
  Week 6 (Day 42): Almost clear | 17
  Week 6 (Day 42): Mild | 5
  Week 6 (Day 42): Moderate | 2
  Week 6 (Day 42): Severe | 0
  Week 6 (Day 42): Very severe | 0
  Week 8 (Day 56): number analyzed (Participants) | 28
  Week 8 (Day 56): Clear | 7
  Week 8 (Day 56): Almost clear | 12
  Week 8 (Day 56): Mild | 7
  Week 8 (Day 56): Moderate | 2
  Week 8 (Day 56): Severe | 0
  Week 8 (Day 56): Very severe | 0
  End of Treatment (last value recorded): Clear | 10
  End of Treatment (last value recorded): Almost clear | 13
  End of Treatment (last value recorded): Mild | 7
  End of Treatment (last value recorded): Moderate | 2
  End of Treatment (last value recorded): Severe | 1
  End of Treatment (last value recorded): Very severe | 0

ADVERSE EVENTS:
Time Frame: From baseline visit (Day -7 to -3) to Follow-up 1 (end of treatment +14 ± 2) and Follow-up 2 (end of treatment +28 ± 2).
Description: Follow-up 1 was only applicable if an adverse event (AE, serious or non-serious) classified as possibly or probably related to the study medication or not assessable in relation to the study medication was present at the participant's last on-treatment visit. This follow-up had to be performed 14 ±2 days after the participant's last on-treatment visit or until final outcome of the AE was determined, whichever came first.
  Follow-up 2 was only applicable in case of possible HPA axis suppression.
Arm/Group | Calcipotriol Plus Hydrocortisone (LEO 80190)
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 15/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Calcipotriol Plus Hydrocortisone (LEO 80190) (N=33)
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Ear disorder (Ear and labyrinth disorders) | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Application site burning (General disorders) | 1
Application site pruritus (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 3
Otitis externa (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Face injury (Injury, poisoning and procedural complications) | 1
Joint sprain (Injury, poisoning and procedural complications) | 1
Ligament injury (Injury, poisoning and procedural complications) | 1
Gout (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Company acknowledges the investigators' right to publish the entire results of the study, irrespective of outcome. The Company retains the right to have any publication submitted to the Company for review at least 30 days prior to the same paper being submitted for publication or presentation. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.